CLINICAL TRIAL: NCT03103321
Title: Testing Decision Aids to Improve Prostate Cancer Decisions for Minority Men
Brief Title: Decision Aids in Improving Knowledge in Patients With Newly Diagnosed Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A191402CD; NCI-2017-00482 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Stage II Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage I Prostate Cancer; PSA Level Five to Ten; PSA Level Less Than Five; PSA Level Ten to Fifty
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A ("Knowing your Options", "Prostate Choice") (Experimental): Patients receive decision aids "Knowing your Options" before and "Prostate Choice" during their consultation visit.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Other: Laboratory Biomarker Analysis
- Arm B ("Knowing your Options") (Experimental): Patients receive "Knowing your Options" decision aid before their consultation visit.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Other: Laboratory Biomarker Analysis
- Arm C ("Prostate Choice") (Experimental): Patients receive "Prostate Choice" decision aid during their consultation visit.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Other: Laboratory Biomarker Analysis
- Arm D (usual care) (Active Comparator): Patients undergo usual care.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Survey Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Internet-Based Intervention — Receive "Knowing your Options" decision aid
  Arms: Arm A ("Knowing your Options", "Prostate Choice"); Arm B ("Knowing your Options")
Other: Internet-Based Intervention — Receive "Prostate Choice" decision aid
  Arms: Arm A ("Knowing your Options", "Prostate Choice"); Arm C ("Prostate Choice")
Other: Best Practice — Undergo usual care
  Other Names: standard of care; standard therapy
  Arms: Arm D (usual care)
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase III trial studies how well decision aids work in improving knowledge in patients with newly diagnosed prostate cancer. Decision aids may improve patients' knowledge of their condition and options for treatment, and may also help when talking with their doctor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the comparative effectiveness of decision aids (DA's) on patient knowledge.

SECONDARY OBJECTIVES:

I. To test the impact of in-visit DA's alone compared to usual care on quality of life outcomes and treatment utilization.

II. To test the impact of out-of-visit DA's alone compared to usual care on quality of life outcomes and treatment utilization.

III. To test the impact of combined in-visit and out-of-visit DA's compared to both usual care and individual DAs on quality of life outcomes and treatment utilization.

IV. To test the comparative effectiveness of DA's on minority men's knowledge. V. To compare clinic time required to administer the DA's across arms.

OUTLINE: Patients are randomized into 1 of 4 arms.

ARM A: Patients receive decision aids "Knowing your Options" before and "Prostate Choice" during their consultation visit.

ARM B: Patients receive "Knowing your Options" decision aid before their consultation visit.

ARM C: Patients receive "Prostate Choice" decision aid during their consultation visit.

ARM D: Patients undergo usual care.

After completion of study, patients are followed up at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have prostate biopsy within 4 months prior to registration showing newly diagnosed prostate cancer, stage T1-3N0M0; in addition, patients must have: Gleason score 6-10
* Prostate-specific antigen (PSA) < 50 ng/mL
* Patients who have had a history of non-cutaneous malignancy in the previous 5 years are not eligible; exception: patients with history of non-melanoma skin cancer are eligible
* Scheduled prostate cancer consultation to be the first consultation after diagnosis (i.e. not a second-opinion or a consultation following previous discussions of treatment options)
* Patients may not be concurrently enrolled to another clinical trial for the treatment of cancer; co-enrollment to biospecimen studies is allowed
* Patients with impaired decision-making capacity (such as with a diagnosis of dementia or memory loss) are not eligible for this study
* Patients must be able to read and comprehend English; non-English-speaking patients may participate so long as an interpreter (e.g., family member, clinic staff, etc.) is present for consent, for the decision aid administration, and gathering of baseline and follow-up measures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2020-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: tilburt.jon@mayo.edu tilburt.jon@mayo.edu, MD, Study Chair — Mayo Clinic
Locations (28):
- United States (28):
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Augusta University Medical Center, Augusta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in the publication PubMed ID 34890060.
Time Frame: The data underlying the publication is available as of and will be available for the duration of the NCTN/NCORP Data Archive.
Access Criteria: Instructions
  1. Click to open the Protocol Section.
  2. Click Edit next to the IPD Sharing Statement and select options for "Plan to Share IPD".
  3. Click Edit next to the References section.
  4. Under the References section, edit the following fields:
     1. Links: https://nctn-data-archive.nci.nih.gov/
     2. Available IPD/Information: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- [Derived] Tilburt JC, Zahrieh D, Pacyna JE, Petereit DG, Kaur JS, Rapkin BD, Grubb RL 3rd, Chang GJ, Morris MJ, Kovac EZ, Babaian KN, Sloan JA, Basch EM, Peil ES, Dueck AC, Novotny PJ, Paskett ED, Buckner JC, Joyce DD, Montori VM, Frosch DL, Volk RJ, Kim SP. Decision aids for localized prostate cancer in diverse minority men: Primary outcome results from a multicenter cancer care delivery trial (Alliance A191402CD). Cancer. 2022 Mar 15;128(6):1242-1251. doi: 10.1002/cncr.34062. Epub 2021 Dec 10. PMID 34890060
- [Derived] Pacyna JE, Kim S, Yost K, Sedlacek H, Petereit D, Kaur J, Rapkin B, Grubb R, Paskett E, Chang GJ, Sloan J, Basch E, Major B, Novotny P, Taylor J, Buckner J, Parsons JK, Morris M, Tilburt JC. The comparative effectiveness of decision aids in diverse populations with early stage prostate cancer: a study protocol for a cluster-randomized controlled trial in the NCI Community Oncology Research Program (NCORP), Alliance A191402CD. BMC Cancer. 2018 Aug 6;18(1):788. doi: 10.1186/s12885-018-4672-3. PMID 30081846

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre- and During-consultation Decision Aids: Patients receive decision aids "Knowing your Options" before and "Prostate Choice" during their consultation visit.
  Internet-Based Intervention: Receive "Knowing your Options" decision aid
  Internet-Based Intervention: Receive "Prostate Choice" decision aid
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Survey Administration: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
- Pre-consultation Decision Aids Only: Patients receive "Knowing your Options" decision aid before their consultation visit.
  Internet-Based Intervention: Receive "Knowing your Options" decision aid
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Survey Administration: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
- During-consultation Decision Aids Only: Patients receive "Prostate Choice" decision aid during their consultation visit.
  Internet-Based Intervention: Receive "Prostate Choice" decision aid
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Survey Administration: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
- Usual Care: Patients undergo usual care.
  Best Practice: Undergo usual care
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
  Survey Administration: Ancillary studies
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care
Started | 25 | 39 | 44 | 50
Completed | 24 | 38 | 43 | 50
Not Completed | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care | Total
Number analyzed (Participants) | 25 | 39 | 44 | 50 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (7.33) | 63.1 (8.09) | 64.6 (7.46) | 63.4 (7.87) | 63.5 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 25 | 39 | 44 | 50 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 25 | 37 | 38 | 47 | 147
  Unknown or Not Reported | 0 | 1 | 4 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Assessed by Prostate Cancer Treatment Questionnaire
Description: The primary outcome, knowledge, will be assessed by a standardized questionnaire (i.e., Prostate Cancer Treatment Questionnaire) administered once, immediately after the clinical consultation while the patient is still at the study site. The number correct from this 12-item measure will be reduced to a percentage of total number correct. With 100%(12 out of 12 item average) being the best possible outcome and 0%(0 out of 12 item average) the worst possible outcome
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of items correct
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care
Number analyzed (Participants) | 24 | 38 | 43 | 50
percentage of items correct | 0.69 (0.165) | 0.65 (0.164) | 0.58 (0.167) | 0.56 (0.232)

2. Secondary Outcome: Decisional Quality as Measured by Decisional Conflict Scale Decisional Regret
Description: The Decisional Regret Scale is a short, 5-item scale measuring "distress or remorse after a (health care) decision." The instrument has been validated in other decision aid studies. Questions are answered on a 5-point agreement scale. A score of 0 means no decisional regret and 5 is the maximum level of regret. The median scores for each cohort were grouped into two categories, 0(no regret) and 1+(at least some regret).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care
Number analyzed (Participants) | 24 | 38 | 43 | 50
Participants
  DCS Total Score of 0 | 13 | 15 | 25 | 30
  DCS Total Score of 1+ | 11 | 23 | 18 | 20

3. Secondary Outcome: Clinical Time Required
Description: Will be compared across DA types using linear mixed models. In particular, this model will include fixed effects for Prostate Choice and Knowing Your Options and a random, site-specific intercept to allow for subjects within the same site to be correlated. Will explore whether the overall effects of interventions on patient knowledge, quality of life, and treatment utilization differ by racial/ethnic subgroups.
Time Frame: 12 months
Measure: Median (Full Range); unit: Minutes
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care
Number analyzed (Participants) | 25 | 39 | 32 | 50
Minutes | 27 [17 to 48] | 38 [13 to 150] | 52.5 [20 to 116] | 39.5 [13 to 250]

4. Secondary Outcome: Quality of Life Assessed by Questionnaire
Description: The Expanded Prostate Cancer Index Composite(EPIC-26) measures health-related quality of life and returns summary scores for urinary, bowel, sexual, and hormonal domains with high test-retest reliability and internal consistency. Scores will be converted into continuous summary scores using standard algorithms. For the EPIC-26 questionnaire, scores were transformed into 0 to 100 scales, with a score of 0 representing the worst possible health-related quality of life and a score of 100 representing the most favorable health-related quality of life. The questionnaire will be administered once; 12 months after the patient's initial consultation.
Time Frame: 12 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care
Number analyzed (Participants) | 25 | 39 | 44 | 50
score on a scale
  Urinary Irritative | 90.63 [68.75 to 100] | 93.75 [56.25 to 100] | 90.63 [43.75 to 100] | 87.5 [37.5 to 100]
  Urinary Incontinence | 96.88 [46 to 100] | 85.5 [14.5 to 100] | 85.5 [8.25 to 100] | 93.75 [8.25 to 100]
  Bowel | 100 [60 to 100] | 100 [70.83 to 100] | 100 [58.33 to 100] | 100 [58.33 to 100]
  Sexual | 33.33 [0 to 95.83] | 36.17 [0 to 100] | 95 [35 to 100] | 90 [35 to 100]
  Hormonal | 92.5 [55 to 100] | 95 [55 to 100] | 95 [35 to 100] | 90 [35 to 100]

5. Secondary Outcome: Utilization as Determined by Chart Review
Description: Will be categorized by the type of treatment the patient received. Will be compared across DA types using linear mixed models. In particular, this model will include fixed effects for Prostate Choice and Knowing Your Options and a random, site-specific intercept to allow for subjects within the same site to be correlated. Will explore whether the overall effects of interventions on patient knowledge, quality of life, and treatment utilization differ by racial/ethnic subgroups.
Time Frame: 12 months
Population: Only includes eligible patients that reached 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care
Number analyzed (Participants) | 16 | 38 | 44 | 50
Participants
  Active surveillance | 4 | 9 | 15 | 16
  Surgery (without radiation) | 6 | 17 | 7 | 12
  Radiation (without surgery) | 5 | 5 | 10 | 18
  Radiation + Surgery | 0 | 0 | 0 | 2
  Treatment Choice Not Listed | 0 | 2 | 6 | 0
  No Treatment (patients that submitted a month 12 form and said No to receiving treatment) | 1 | 5 | 6 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Description: This study did not collect adverse events.
  We do not anticipate any additional adverse events related to participation in this study beyond usual care. If patients experience any emotional discomfort when completing the questionnaires, they may choose not to complete them and/or speak with the site staff. Patients experiencing any physical or psychological complications related to their standard of care treatment should discuss this with their treating physician.
Arm/Group | Pre- and During-consultation Decision Aids | Pre-consultation Decision Aids Only | During-consultation Decision Aids Only | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/38 | 1/43 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT03103321/Prot_SAP_000.pdf